CLINICAL TRIAL: NCT00927979
Title: Phase 3 Prospective, Randomized, Controlled and Double-blinded Second Trial on Pain Relief by Continuous Intra-peritoneal Nebulization of Ropivacaine Under Remifentanil Anesthesia, During Gynecological Laparoscopic Surgery
Brief Title: Pain Relief by Intra-Peritoneal Nebulization of Ropivacaine Under Remifentanil Anesthesia for Gynecological Laparoscopy
Acronym: PSDR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Ostrovsky Ludmila, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMC090074CTIL; PSDR (Other: Gynecology Dept. Code)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Gynecological Laparoscopy
MeSH Terms: interventions — Water; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Experimental)
  Interventions: Drug: 10 mLRopivacaine 1%; Drug: 10 mL Ropivacaine 1%
- Water for injection (Placebo Comparator)
  Interventions: Drug: Water for injection

INTERVENTIONS:
Drug: 10 mLRopivacaine 1% — Intraperitoneal nebulization of 10 mL Ropivacaine 1%
  Arms: Ropivacaine
Drug: Water for injection — Intraperitoneal nebulization of 10 mL water for injection
  Arms: Water for injection
Drug: 10 mL Ropivacaine 1% — Intraperitoneal nebulization of 10 mL Ropivacaine 1%
  Arms: Ropivacaine

SUMMARY:
In our prospective, randomized, placebo controlled and double-blinded study we will study the efficacy of intraperitoneal ropivacaine nebulization on pain relief during gynecologic laparoscopic surgery. This is a second steady with protocol of general anesthesia used of Remifentanil.

DETAILED DESCRIPTION:
Outcome Measures :

* VAS score
* Use of analgesics during operation and postoperative period

ELIGIBILITY:
Inclusion Criteria:

* Elective gynecological laparoscopic surgery including unilateral or bilateral salpingo-oophorectomy or ovarian cystectomy
* Patient not participating in other medical study at present or during the last 30 days
* Patient is capable of reading, understanding and signing on an informed consent
* Age 18 years and above
* ASA physical status grade 1-2

Exclusion Criteria:

* Allergy to ropivacaine or other local anesthetics or other medications listed in the protocol
* Acute pelvic inflammatory disease
* Coumadin or aspirin treatment
* Significant arrythmias
* Analgesic treatment for chronic pain
* BMI>35

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score (VAS) | 24 hours

SECONDARY OUTCOMES:
Use of Analgesics | 24 hours